CLINICAL TRIAL: NCT05498207
Title: Identification of Biomarkers for Stress Vulnerability and Resilience
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Pritzker Consortium (Other); Weill Medical College of Cornell University (Other); Hope for Depression Research Foundation (Other)
Responsible Party: Principal Investigator, Huda Akil, Professor of Neurosciences, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00211856
Record Dates: First submitted 2022-08-09; First posted 2022-08-11 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Healthy
Keywords: Mental Health; Mobile application; Cognitive Behavioral Therapy (CBT); Stress; Fitbit
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Participants that have a Android will be assigned to the no intervention arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No Intervention (No Intervention): Participants will complete assessments at baseline, 3 months, 6 months, 9 months and 12 months. (this includes specimen collections, interviews, and surveys). Participants will also be asked to wear a Fitbit for 12 months.
- Maya mobile app (Experimental): Maya mobile app- CBT based self-help app
  Interventions: Behavioral: Maya App

INTERVENTIONS:
Behavioral: Maya App — Participants will utilize the Maya App for at least 20 minutes per day, 2 days per week, for 6 weeks. Additionally, participants will complete assessments at baseline, 3 months, 6 months, 9 months and 12 months (this includes specimen collections, interviews, and surveys). Participants will also be asked to wear a Fitbit for 12 months.
  Arms: Maya mobile app

SUMMARY:
The purpose of this research study is to understand the biological mechanisms of stress vulnerability (being susceptible to stress) and stress resilience (being able to recover readily from stress), obtain biomarkers (a biological indicator) for stress resilience and to devise strategies for prevention and treatment of stress-related disorders.

DETAILED DESCRIPTION:
This study will be using the Maya application (app) for the intervention arm, a mobile cognitive behavior therapy (CBT) program for adolescents and young adults experiencing anxiety symptoms. The Maya app, developed at Weill Cornell, teaches cognitive behavioral therapy (CBT) techniques including emotion monitoring, cognitive restructuring, mindfulness, and exposure to help individuals with anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Incoming Freshmen Students at the University of Michigan

Exclusion Criteria:

* Suicidal Ideation

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-23 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety symptoms based on the General Anxiety Disorder-7 Scale (GAD-7) between the intervention arm and the no intervention arm | Baseline, up to 12 months
  The GAD-7 is a 7 item questionnaire to measure the severity of anxiety symptoms (scores between 0-21). The items measure both psychic anxiety and somatic anxiety, where higher scores, defined by a score range of greater than or equal to 10, indicate a greater presence of symptoms and lower scores, defined by a score range of 0-9, indicate mild to no anxiety symptoms. Change in anxiety ratings between the intervention arm and the no intervention arm.
Change in depressive symptoms based on the Patient Health Questionnaire-9 (PHQ-9) between the intervention arm and the no intervention arm | Baseline, up to 12 months
  The PHQ-9 is a 9-item scale containing three subscales measuring physical, cognitive, and social concerns regarding depression. Higher scores, defined by a score range of greater than or equal to 10, reflect greater presence of symptoms and lower scores, defined by a score range of 0-9, indicate mild to no depression symptoms. Change in depression ratings between the intervention arm and the no intervention arm.
Change in anxiety symptoms based on the Spielberger State and Trait Anxiety Inventory (STAI) between the intervention arm and the no intervention arm | Baseline, up to 12 months
  The Spielberger State and Trait Anxiety Inventory is a validated self-reporting instrument used to assess anxiety. The inventory consists of state anxiety, which evaluates how the subject feels currently (transient anxiety) and trait anxiety (anxiety related to personality). The scale consists of 20 questions to determine state and 20 questions for trait anxiety with a 4-point Likert scale, a higher score indicates greater anxiety. Total score for state and trait measures ranges from 20 (no anxiety) to 80 (maximum anxiety). Change in anxiety ratings between the intervention arm and the no intervention arm.

CONTACTS AND LOCATIONS:
Overall Officials: Huda Akil, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of the proposed study will be shared with the scientific community after deidentification. The analytic code the team used will also be shared. Sharing will require a proposal from scientists who specify the questions to be asked and describe methodologically sound approaches to address their aims. Proposals should be directed to akil@umich.edu. To get access to the data, requestors will need to sign a data transfer and use agreement.
Supporting Information: ICF
Time Frame: Data will be made available upon full publication of the results and will end 36 months following article publication.